CLINICAL TRIAL: NCT04148183
Title: Randomized Clinical Trial, Effect of Metformin and Rosiglitazone Over Glucose Homeoastasis in no Diabetic With Metabolic Syndrome Patients.
Brief Title: Effect of Metformin and Rosiglitazone Over no Diabetic With Metabolic Syndrome Patients.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: J JESUS VENEGAS, MD (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); National Council of Science and Technology, Mexico (Other)
Responsible Party: Sponsor-Investigator, J JESUS VENEGAS, MD, Master Degree, Nephrologist, Universidad de Colima
Organization: Universidad de Colima (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ucol-1
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Metformin; Rosiglitazone; Control Groups

STUDY DESIGN:
Intervention Model Description: Prior to detailed information and signature of informed consent by patients, it was randomized forming three treatment groups, a) Placebo, b) Metformin (850 mg/day), c) Rosiglitazone (4 mg/day), treatment was administered for 8 weeks
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin Group (Experimental): Metformin (850 mg/day) treatment was administered for 8 weeks
  Interventions: Drug: Metformin group
- Rosiglitazone Group (Experimental): Rosiglitazone (4 mg/day), treatment was administered for 8 weeks
  Interventions: Drug: Rosiglitazone group
- Placebo Group (Placebo Comparator): Placebo treatment was administered for 8 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metformin group — We add treatment with Metformin (850 mg/day), treatment was administered for 8 weeks
  Other Names: Metformina
  Arms: Metformin Group
Drug: Rosiglitazone group — we add Rosiglitazone (4 mg/day), treatment was administered for 8 weeks
  Other Names: Rosiglitazona
  Arms: Rosiglitazone Group
Drug: Placebo oral tablet — We add Placebo, treatment was administered for 8 weeks
  Other Names: Control Group
  Arms: Placebo Group

SUMMARY:
To compare the effect of insulin sensitizing drugs (metformin and rosiglitazone) over glucose homeostasis (GH) in no diabetic metabolic syndrome individuals. A randomized blinded clinical trial did in patients with metabolic syndrome (n=30), without diabetes. Prior to detailed information and signature of informed consent by patients were done three treatment groups by randomized technique; a) Placebo, b) Metformin (850 mg/day), c) Rosiglitazone (4 mg/day), treatment was administered for 8 weeks. GH was measured before and after treatment using oral glucose tolerance test (OGTT), and IR-index (Homeostatic Model). Determination was performed on weight, size, body mass index, plicometry, blood pressure, fasting glucose levels, triglycerides, HDL-cholesterol and insulin.

DETAILED DESCRIPTION:
Metabolic syndrome is a risk factor for diabetes mellitus characterized by insulin resistance, hypertension, triglyceride elevation, low levels of high-density lipoproteins, and obesity. Metformin and rosiglitazone are two insulinosensensitizers used in the treatment of diabetes. Now there is controversy over the use of insulinossensitizers in non-diabetic patients with metabolic syndrome. To compare the effect of insulin sensitizing drugs (metformin and rosiglitazone) over glucose homeostasis (GH) in no diabetic metabolic syndrome individuals. Randomized blinded clinical trial in patients with metabolic syndrome without diabetes was done, sample size (n=30). Prior to detailed information and signature of informed consent by patients was randomized forming three treatment groups, a) Placebo, b) Metformin (850 mg/day), c) Rosiglitazone (4 mg/day), treatment was administered for 8 weeks. GH was measured before and after treatment using oral glucose tolerance test (OGTT), and IR-index (Homeostatic Model). Determination was performed on weight, size, body mass index, plicometry, blood pressure, fasting glucose levels, triglycerides, HDL-cholesterol and insulin. Statistic no parametric (Kruskal Wallis, Wilcoxon, U Mann Whitney) to compare characteristics inter o intra groups was done. Exact Fisher test was used for qualitative variable, and consider significance with p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old.
* Metabolic Syndrome criteria of World Health Organization .

Exclusion Criteria:

* Diabetes Mellitus
* Allergic to Metformin,
* Allergic to rosiglitazone.
* Hepatic disease.
* Hearth disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2005-01-01 (Actual); Study Completion 2009-01-01 (Actual)

PRIMARY OUTCOMES:
INSULIN RESISTANCE | 8 weeks
  INSULIN RESISTANCE index (Homeostatic Model) is method that need insulin concentration and glucose in blood to calculate index.

SECONDARY OUTCOMES:
oral glucose tolerance test (OGTT), | 8 weeks
  oral glucose tolerance test was done take a sample of blood before a period without feed of 8 hours, we took a blood glucose sample then we gave a 75g of glucose and after we took blood glucose at the hour and 2 hours of OGTT test

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Tene, DS, Study Director — Universidad de Colima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seufert J, Lubben G, Dietrich K, Bates PC. A comparison of the effects of thiazolidinediones and metformin on metabolic control in patients with type 2 diabetes mellitus. Clin Ther. 2004 Jun;26(6):805-18. doi: 10.1016/s0149-2918(04)90125-7. PMID 15262452
- [Background] Gulias-Herrero A, Aguilar-Salinas CA, Gomez-Perez FJ, Rull JA. The combination metformin/glyburide exerts its hypoglycemic effect mainly by increasing insulin secretion: a controlled, randomized, double-blind, crossover study. Diabetes Nutr Metab. 2003 Oct-Dec;16(5-6):268-76. PMID 15000437
- [Background] Davidson MB. Is treatment of insulin resistance beneficial independent of glycemia? Diabetes Care. 2003 Nov;26(11):3184-6. doi: 10.2337/diacare.26.11.3184. No abstract available. PMID 14578261
- [Background] Lehtovirta M, Forsen B, Gullstrom M, Haggblom M, Eriksson JG, Taskinen MR, Groop L. Metabolic effects of metformin in patients with impaired glucose tolerance. Diabet Med. 2001 Jul;18(7):578-83. doi: 10.1046/j.1464-5491.2001.00539.x. PMID 11553189
- [Background] Derosa G, D'Angelo A, Ragonesi PD, Ciccarelli L, Piccinni MN, Pricolo F, Salvadeo SA, Montagna L, Gravina A, Ferrari I, Paniga S, Cicero AF. Metabolic effects of pioglitazone and rosiglitazone in patients with diabetes and metabolic syndrome treated with metformin. Intern Med J. 2007 Feb;37(2):79-86. doi: 10.1111/j.1445-5994.2007.01238.x. PMID 17229249
- [Background] Mohiyiddeen L, Watson AJ, Apostolopoulos NV, Berry R, Alexandraki KI, Jude EB. Effects of low-dose metformin and rosiglitazone on biochemical, clinical, metabolic and biophysical outcomes in polycystic ovary syndrome. J Obstet Gynaecol. 2013 Feb;33(2):165-70. doi: 10.3109/01443615.2012.745839. PMID 23445141